CLINICAL TRIAL: NCT07014020
Title: An Open-label, Single Arm, Dose-Escalation Clinical Study to Evaluating the Safety, Tolerability and Preliminary Efficacy of a Single Intracerebroventricular Injection of RB001 for the Treatment of SHANK3-related Phelan McDermid Syndrome.
Brief Title: RB001 Gene Therapy Study in Children With SHANK3-related Phelan McDermid Syndrome (PMS)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Shenzhen Reborngene Therapeutics Co., Ltd. (Unknown); Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, Ye Wu, Professor, Chief Physician, Peking University First Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RB001-101; 2025R0116-0002 (Other: EC of Peking UFH)
Record Dates: First submitted 2025-05-21; First posted 2025-06-10 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-06

CONDITIONS: Phelan-McDermid Syndrome; SHANK3 Haploinsufficiency
Keywords: AAV; SHANK3; Phelan-Mecdermid Syndrome; 22q13.3 deletion syndrome
MeSH Terms: conditions — Telomeric 22q13 Monosomy Syndrome

STUDY DESIGN:
Intervention Model Description: An Open-label, Single Arm, Dose-Escalation Clinical Study to Evaluating the Safety, Tolerability and Preliminary Efficacy of a Single Intracerebroventricular Injection of RB001
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RB001 (Experimental): Once intracerebroventricular injection; The duration of the study is about 14 months for each subject, including a 2-month screening period, an inpatient period from Day 1 (Dosing) to Day 7 post-administration and a subsequent 12-month outpatient follow-up period.
  Interventions: Genetic: RB001

INTERVENTIONS:
Genetic: RB001 — The study will enroll up to 2 cohorts, evaluating a starting dose plus a higher or lower dose

SUMMARY:
This is a first in human, open-label, dose-escalation study to evaluate the safety, tolerability, and clinical activity of a single dose of RB001 administered via intracerebroventricular (ICV) injection in pediatric with SHANK3 related Phelan-McDermid Syndrome. Clinical data will be evaluated for safety, tolerability, and preliminary efficacy of RB001 in participants with SHANK3 related PMS.

DETAILED DESCRIPTION:
SHANK3-related Phelan McDermid syndrome (PMS) is a rare neurodevelopmental disorder primarily caused by a deletion of chromosome 22q13 or a mutation of the SHANK3 gene. The syndrome is characterized by intellectual disability and language impairment. The SHANK3 protein is part of the postsynaptic density complex and participates in postsynaptic signal transduction and synaptic development, serving as a critical structural protein for central nervous system development and functional maintenance. SHANK3 deficiency leads to abnormal neuronal development and is the primary cause of PMS. The estimated global prevalence is approximately 1/15,000. Clinical manifestations include global developmental delay, particularly severe language delay, autism-like behaviors, hypotonia, and potentially epilepsy. Currently, there are no effective treatments for this condition.

RB001 is developed by Shenzhen Reborngene Therapeutics Co., Ltd. for the treating of Phelan-McDermid Syndrome. RB001 utilizes the Adeno-Associated Virus (AAV) vector to deliver an optimized SHANK3-minigene via intracerebroventricular (ICV) injection. Nonclinical studies have demonstrated that a single ICV injection of RB001 could restore SHANK3 mRNA and protein expression in the target region of central nervous system of the SHANK3-mutant mouse models, as well as the restore of motor deficits, stereotypical behaviors, and reduced exploratory behaviors and neuronal function.

A target of 8 pediatric participants aged 3 to 18 years will be treated. All participants will be followed for safety, tolerability and preliminary efficacy after the date of treatment with RB001.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥3 years and <18 years (at the time of signing informed consent), any gender
* Genetic test and clinical confirmed diagnosis of SHANK3-related PMS
* Meets diagnostic criteria for moderate or more severe Autism Spectrum Disorder (ASD)
* Intelligence Quotient (IQ) score <70 or Developmental Quotient (DQ) (excluding gross motor) average score <70
* Willing to provide biological samples required for the study (e.g., blood, urine)
* Consent to hospitalization for intracerebroventricular injection surgery
* The holders of parental authority who are able to understand and willing to comply with study requirements and procedures, voluntarily participating and signing the informed consent

Exclusion Criteria:

A pediatric participant who meets any of the following criteria will be excluded from this study:

* Previous or current participation in other PMS drug clinical trials or other AAV gene therapy clinical studies
* Has known allergic constitution, including allergy or hypersensitivity to prednisone acetate, other glucocorticosteroids, their excipients, or local anesthetics
* Subjects with status epilepticus within 3 months prior to enrollment
* Subjects requiring invasive or non-invasive ventilatory support
* Serum anti-AAV neutralizing antibody titer >1:200
* Significant laboratory abnormalities: alanine aminotransferase (ALT), aspartate aminotransferase (AST), γ-glutamyl transferase (GGT) with any value above the upper limit of normal; total bilirubin above the upper limit of normal; creatinine ≥159 μmol/L; hemoglobin (Hb) <80 g/L; prothrombin time (PT) prolonged by ≥3 seconds; activated partial thromboplastin time (APTT) prolonged by ≥10 seconds; fasting blood glucose ≥7.0 mmol/L; glycated hemoglobin (HbA1c) ≥6.5%; platelets (PLT) <100×10^9/L
* Subjects with liver disease or history of heart disease that may pose drug-related risks as assessed by the investigator
* Subjects deemed unsuitable for intracerebroventricular administration or with other special circumstances as assessed by the investigator
* Positive for human immunodeficiency virus antibody, hepatitis B surface antigen, hepatitis C antibody, syphilis antibody, active TORCH virus infection, or active Epstein-Barr virus infection
* Concomitant use of any of the following medications within 90 days prior to administration, or planned immunosuppressive treatment within 3 months after starting the trial, except for prophylactic medications specified in the protocol (cyclosporine, tacrolimus, methotrexate, cyclophosphamide, intravenous immunoglobulin, rituximab, etc. )
* Other conditions deemed unsuitable for participation in this study by the investigator

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  Types, severity, and incidence of adverse events (AEs) and serious adverse events (SAEs) within 52 weeks after RB001 injection

SECONDARY OUTCOMES:
To evaluate the changes on Clinical Global Impression Scale - Severity (CGI-S) after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes from baseline at weeks 12, 26, and 52 after RB001 injection.
  Clinical Global Impression Scale (CGI) severity item provided with a seven-point scale of severity of patient's clinical condition (1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.)
To evaluate the changes on Clinical Global Impression Scale - Improvement (CGI-I) after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes from baseline at weeks 12, 26, and 52 after RB001 injection.
  Clinical Global Impression Scale (CGI) Improvement item provided with a seven-point scale of improvement of patient's clinical condition (1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment.)
To evaluate the changes on Patient's Global Impressions of Improvement (PGI-I) after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes from baseline at weeks 12, 26, and 52 after RB001 injection.
  The PGI-Improvement scale is a transition scale that is a single question asking the patient to rate their urinary tract condition as compared with how it was prior to before beginning RB001 injection on a scale from 1. Very much better to 7. Very much worse
To evaluate the changes on Childhood Autism Rating Scale (CARS-2) after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes from baseline at weeks 12, 26, and 52 after RB001 injection.
  In the CARS-2, the rater observes the behavior of the child in specific situations and assigns scores based on a series of 15 descriptive items (including: Relating to People, Imitation, Emotional Response, Body Use, Object Use, Adaptation to Change, etc.). Each item is scored on a range of 0 to 4, with 0 indicating no abnormality and 4 indicating severe abnormality. The rater also considers the overall impression and severity of the child, resulting in a total score. The total score falls between 15 and 60, with higher scores indicating a higher level of autism severity.
To evaluate the changes on Autism Behavior Checklist (ABC) after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes from baseline at weeks 12, 26, and 52 after RB001 injection. In the Autsim Autism Behavior Checklist (ABC), the rater (usually the Guardian) observes the child's behavior and score 57 specific items across five domains (Sensory Behavior, Relating Behavior, Body and Object Use, Language, and Social/Self-Help). Each item is rated 1-4 based on behavior frequency/severity (1=absent, 4=severe). The total score (57-228) is calculated, with higher scores indicating greater autism-related behavioral impairment. A score ≥53 suggests clinical concern for autism spectrum disorder.
To evaluate the changes on Griffith developmental assessment scale - Chinese (GDS-C) after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes of developmental trajectories from baseline at weeks 12, 26, and 52 after RB001 injection, the Griffiths Developmental Assessment Scale - Chinese Version (GDS-C) is accessed by certified examiners. The scale evaluates 240 age-standardized tasks across six domains (Locomotor, Personal-Social, Language, Eye-Hand Coordination, Performance, and Practical Reasoning). Tasks are scored 0 or 1 (1=pass, 0=fail), with raw scores converted to Developmental Quotients (DQ) using China-specific norms (2020 revision). DQ<85 suggests potential mild developmental delay, while a multi-domain DQ<70 indicates significant developmental delay.
To evaluate the changes on Wechsler Preschool and Primary Scale of Intelligence (WPPSI) or Wechsler Intelligence Scale for Children (WISC) after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate cognitive changes from baseline at weeks 12, 26, and 52 after RB001 injection, the Wechsler Intelligence Scales are administered based on baseline age: WPPSI for subjects aged 2.5-7.7 years at screening, WISC for subjects aged 6-16 years at screening.
  the certified neuropsychologist conducts assessments under standardized conditions and assigns scores based on five scales (Verbal Comprehension, Visual Spatial, Fluid/Quantitative Reasoning, Working Memory, Processing Speed) to derive a Full Scale IQ. Scores are norm-referenced (mean=100, SD=15), with higher values indicating superior cognitive ability. IQ<85 suggests potential mild cognitive delay, while IQ<70 indicates significant cognitive delay.
To evaluate the changes on Adaptive Behavior Assessment System-Second Edition (ABAS-2) after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes of functional adaptive behaviors from baseline at weeks 12, 26, and 52 after RB001 injection, the Adaptive Behavior Assessment System-Second Edition (ABAS-2) is administered. the rater (usually the Guardian) score the child's daily living skills across 10 domains (Communication, Self-Care, Social, etc.) using age-specific questionnaires. Items are scored 0-3 based on frequency of competent performance, and raw scores normalized to standard scores based on ages (mean=100, SD=15). The General Adaptive Composite (GAC) serves as the primary secondary endpoint. CAG < 85 suggests potential mild delay, while CAG ≤ 70 indicates significant delay.
To evaluate the changes on Social Life Ability Scale For Infant-Junior Middle School Student (S-M) after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate adaptive functioning from baseline at weeks 12, 26, and 52 after RB001 injection, the Social Life Ability Scale for Infants-Junior Middle School Students (S-M Scale) is administered. Parents or primary caregivers observe the child's daily behaviors and score 132 specific items across six functional domains (Independent Living Skills, Motor Abilities, Practical Task Performance, Communication Skills, Self-Management, and Socialization). Each item is scored 0 or 1 (1 = pass, 0 = fail) based on observed capability. The total score (0-132) is calculated by summing all items, with higher scores indicating better adaptive functioning. A standard score ≤9 (equivalent to a raw score ≤70; ≥2 SD below the norm) suggests significant impairment in social adaptive abilities.
To evaluate the changes on Child Behavior Checklist (CBCL) after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate behavioral/emotional problems from baseline at weeks 12, 26, and 52 after RB001 injection, the Child Behavior Checklist (CBCL) is administered. Parents or caregivers rate the child's behaviors using 113+ problem items across empirically based syndromes (Anxious/Depressed, Withdrawn/Depressed, Somatic Complaints, Social Problems, Thought Problems, Attention Problems, Rule-Breaking Behavior, and Aggressive Behavior). Each item is scored 0-2 (0 = not true, 1 = somewhat/sometimes true, 2 = very/often true). The total problem score (0-240) is calculated by summing all items, with higher scores indicating greater behavioral/emotional impairment. A T-score >63 (>90th percentile) suggests clinical concern, and >70 (>98th percentile) indicates. (T-scores (M = 50, SD = 10) are derived from normative samples)
To evaluate AAV viral load after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate viral load dynamics from baseline, at Day 7, Weeks 4, 8, 12, 26, and 52 after RB001 injection, blood samples will be collected at each time point. Viral load will be quantified using RT-qPCR. (Sampling will be discontinued if viral load falls below the lower limit of detection for three consecutive measurements.)
To evaluate AAV viral shedding after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate Viral shedding from baseline, and at Day 7, Weeks 4, 8, 12, 26, 52 after RB001 injection. Saliva, urine, and feces samples will be collected at each time point. Viral load will be quantified using RT-qPCR. (Sampling will be discontinued if viral load falls below the lower limit of detection for three consecutive measurements.)
To evaluate AAV binding and neutralizing antibodies after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate AAV binding and neutralizing antibodies (Abs) dynamics from baseline, and at Day 7, Weeks 4, 8, 12, 26, 52 after RB001 injection. blood samples will be collected at each time point. Antibodies will be quantified using ELISA (for binding Ab) and cell-coculture (for neutralizing Ab). (Sampling will be discontinued if tests results are negative for three consecutive measurements.)
To evaluate SHANK3 binding antibody after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate SHANK3 binding antibody (Ab) dynamics from baseline, and at Weeks 4, 8, 12, 26, 52 after RB001 injection. blood samples will be collected at each time point. Antibodies will be quantified using ELISA. (Sampling will be discontinued if tests results are negative for three consecutive measurements.)
To evaluate changes in T-cell responses against AAV and SHANK3 after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes in T-cell responses against AAV and SHANK3 from baseline and at Weeks 26 and 52 after RB001 injection, blood samples will be collected at each time point. Antigen-specific T-cell responses will be quantified using ELISpot assays with peptide pools spanning AAV capsid and SHANK3 epitopes libraries.

OTHER OUTCOMES:
To evaluate changes in sleep patterns after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes in sleep patterns from baseline at Weeks 12, 26, 52 after RB001 injection. Sleep latency, total wake time, number of awake bouts, total sleep time, sleep onset time, final awakening time, and sleep initiation interventions will be recorded.
To evaluate changes in facial processing and emotional perception abilities after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes in facial processing and emotional perception abilities from baseline at Weeks 12, 26 and 52 after RB001 injection, eye movement patterns will be recorded using programmed eye-tracking equipment (Tobii Pro Fusion) while participants view dynamic emotional faces (happy, fear, neutral) and control house stimuli. Task completion status (especially valid fixation rate) and protocol adherence metrics will be documented.
To evaluate the changes in olfactory performances after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes in olfactory performance from baseline and at Weeks 12, 26 and 52 after RB001 injection. Respiratory rate, duration, ventilation volume in response to five olfactory stimuli will be documented using airflow monitoring and olfactory testing.
  The olfactory stimuli comprised two pleasant fragrant oils (pineapple and chocolate), two unpleasant odor compounds (trimethylamine and isovaleric acid) and blank control (air). Trimethylamine has a rotten fish-like odor and isovaleric acid has a sour stinky foot-like odor.
To evaluate the changes in Electroencephalogram (EEG) patterns after a single intracerebroventricular injection of RB001 through week 52 | 52 weeks
  To evaluate changes in EEG patterns from baseline and at Weeks 12, 26, and 52 following RB001 injection. The power of spectral band (delta, theta, alpha, beta) of EEG will be recorded under four independent conditions: two resting state (eyes closed and eyes open) and two task states (watching cartoon and cartoon without sequence) using a portable EEG system.
To evaluate the effects of higher cognitive functions up to 52 weeks after a single intracerebroventricular administration of RB001 | 52 weeks
  To evaluate changes in higher cognitive functions from baseline and at Weeks 12, 26, and 52 following RB001 injection. Subjects will enter an enriched space equipped with a slide, ball pit balls, foam mats, and various toys. His/her behavior will be recorded for 10 minutes using four corner-mounted cameras. Motion trajectories, stereotypic behaviors, and interactions with different objects (or persons) will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University First Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No